CLINICAL TRIAL: NCT04393103
Title: Role of Intralipid in Management of Organophosphorus Poisoning
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: no avilable resorces
Sponsor: Amani Hassan Abdel-Wahab (Other)
Responsible Party: Sponsor-Investigator, Amani Hassan Abdel-Wahab, Professor of anesthesia and intensive care, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AssiutU_HAA_OP_poisoning
Record Dates: First submitted 2020-04-27; First posted 2020-05-19 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Organophosphorus Poisoning
Keywords: intralipid, organophosphorus poisoning
MeSH Terms: conditions — Organophosphate Poisoning | interventions — soybean oil, phospholipid emulsion; Atropine

STUDY DESIGN:
Intervention Model Description: Atropine will be administered to ALL PATIENTS by doubling dose method which comprised of administering atropine start-ing from 2mg and to double the dose and administer till com-plete atropinization. Following this an infusion of 10-20% of the atropinizing dose was given every hour.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Follow up (Other): Follow Up of 30 patients after administration of atropine.
  Interventions: Drug: Intravenous Atropine Sulfate
- intralipid 20% adjuvant (Experimental): 30 patients will receive atropine and intralipid AS AN ADJUVANT Three boluses of IFE 15 mg/kg were given over 3 minutes, 20 minutes apart.
  Interventions: Drug: Intralipid, 20% Intravenous Emulsion; Drug: Intravenous Atropine Sulfate

INTERVENTIONS:
Drug: Intralipid, 20% Intravenous Emulsion — Atropine will be administered to ALL PATIENTS by doubling dose method which comprised of administering atropine start-ing from 2mg and to double the dose and administer till com-plete atropinization. Following this an infusion of 10-20% of the atropinizing dose was given every hour.
  * Group A (Control Group) : Follow Up of 30 patients.
  * Group B (Study Group): 30 patients will receive intralipid AS AN ADJUVANT Three boluses of IFE 15 mg/kg were given over 3 minutes, 20 minutes apart.
  Other Names: lipofundin 20
  Arms: intralipid 20% adjuvant
Drug: Intravenous Atropine Sulfate — Atropine will be administered to ALL PATIENTS in Group A and group B by doubling dose method which comprised of administering atropine start-ing from 2mg and to double the dose and administer till complete atropinization. Following this, an infusion of 10-20% of the atropinizing dose was given every hour.
  Other Names: Atropine 1 mg / 1 ml

SUMMARY:
Aim of the study:

To assess the role of intralipid emulsion in the acute man-agement of organophosphorus toxicity and its benefits in de-creasing mortality rates among victims.

DETAILED DESCRIPTION:
Organophosphates (OPs) are cholinesterase inhibitors that are widely used as pesticides and organophosphate (OP) poisoning is an important public health concern in Egypt especially in the rural farming population. Organophosphate toxicity lead to a characteristic toxidrome that includes muscarinic, nicotinic and central nervous system signs and symptoms and, without proper and early antidotal treatment, death. A new antidote is the need of the hour. Lipid emulsion being inexpensive, easily available and effective in management of other lipid soluble toxins may be a novel option. The exact mechanisms by which ILE exert their beneficial effects are not fully understood, and several have suggested synergistic effects of several mechanisms. The mechanisms of action can be divided into intravascular, membrane, and intracellular effects. The original theory explaining the mechanism of lipid rescue was that of "lipid sink", suggesting sequestration of lipophilic compounds to an expanded intravascular lipid phase, extracting the offending agent from the target tissue, and reversing the toxicity. Other hypotheses relate to the mechanism by which ILEs facilitate cardiac rescue from drug poisoning. These include:

1. increasing myocardial energy substrate delivery and a direct cardiotonic effect of ILE on the poisoned heart.
2. an effect of ILE on calcium ion channels through high levels of long-chain fatty acids, leading to increased cardiomyocyte calcium and positive inotropic effect.

ELIGIBILITY:
Inclusion Criteria:

* Age group of 18-60 years who are exposed to organophosphorus compounds.
* Clinical manifestations of organophosphorus toxidromes (hyper-salivation, lacrimation, sweating, urinary incontinence, di-arrhea, vomiting and abdominal pain).

Exclusion Criteria:

1. Patient or relative in charge refusal.
2. Chronic renal or liver disease manifested by history, clinical and investigatory diagnosis.
3. Previous history of acute or chronic pancreatitis
4. Combined poisoning with non OP compounds
5. Asymptomatic patients.
6. Contraindications to intralipid emulsion as:

   * disturbances of normal fat metabolism such as patho-logic hyperlipemia manifested by history, clinical and investigatory diagnosis.
   * lipoid nephrosis manifested by history, clinical and investigatory diagnosis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
duration in days of hospitalization and ICU stay | four days
  The primary outcome is to study the difference in total days of hospitalization and ICU stay between the study and control groups.

SECONDARY OUTCOMES:
mortality. | four days
  Death among cases under study.

CONTACTS AND LOCATIONS:
Overall Officials: Hamdy A. Youssef, Professor, Study Director — Professor of anesthesia and intensive care, Assiut University

IPD SHARING:
Plan to Share IPD: No